CLINICAL TRIAL: NCT04241237
Title: Concordance Between Liquid and Tissue Biopsy in Newly Diagnosed Metastatic Breast Cancer
Brief Title: Concordance Between Liquid and Tissue Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Epic Sciences (Industry); University of Western Ontario, Canada (Other); Lunenfeld Tanenbaum Research Institute (Other); MOUNT SINAI HOSPITAL (Other); Toronto Sunnybrook Regional Cancer Centre (Other); University of Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Concordance
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Circulating Tumor Cells; Circulating Tumor DNA; Liquid Biopsy; Tissue biopsy; Concordance
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and archival tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic Breast Cancer patients: Investigators plan to enroll patients who are undergoing biopsy for potential metastatic Breast Cancer any subtype ER/PgR+ and HER2, triple negative or HER2+ at least 6 months before suspected metastases were identified. The suspected metastases in these patients must be outside the ipsilateral breast, axilla infra/supraclavicular areas. In those with suspected metastases in contralateral axilla, infra/supraclavicular areas only a new contralateral breast primary must be excluded by physical exam, mammogram and MRI
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Blood will be drawn from each patient to check the concordance between liquid and tissue biopsy

SUMMARY:
Tissue biopsy is a procedure to remove a piece of tissue (sample of cells) from the body to be analyzed in a laboratory, and it is commonly performed to confirm diagnosis of a patient with symptoms of breast cancer recurrence. It may also provide information on tumor markers (hormone receptors, HER2) that can guide treatment decisions. The goal of this study is to determine whether blood tests (which require less-invasive procedures) can be used to confirm diagnosis of suspected recurrent breast cancer (as compared to tissue biopsy).

Investigators plan to investigate blood factors which include circulating tumor cells (CTCs - i.e., cancer cells that can be detected in the blood), circulating tumor DNA (ctDNA - i.e., pieces of DNA from cancer cells that can be found in the blood), as well as other biomarkers. Investigators will conduct this study in 120 participants who present with suspected breast cancer recurrence and symptoms of cancer that has spread to other areas in the body.

Participants will be asked for blood collection within 30 days before tissue biopsy. The tissue will be analysed locally to determine the presence of cancer and the tumor markers listed above. The blood will be processed and stored for analysis of CTCs and ctDNA. If these blood tests show concordance with tissue based tests (presence of cancer cells, hormone receptors & HER2 status), these tests could be used in future studies to confirm diagnosis using a non-invasive procedure. Also, investigators believe that the results of this study can influence other research of early-stage recurrent breast cancer.

DETAILED DESCRIPTION:
In Canada, it is estimated that more than 26,900 women will be diagnosed with breast cancer (BC), and 5,000 women will die from BC in 2019. Metastatic BC will cause the vast majority of these deaths. Tissue biopsy is recommended to confirm recurrence (presence of cancer cells) in patients with a history of previous BC. Additionally, tissue biopsy provides information on BC subtypes (estrogen receptor (ER), progesterone receptor (PgR), and HER2 status). Technological advances over the last several years have led to more robust methods for the detection, quantification, and characterization of liquid biopsy (including CTCs and ctDNA) in recurrent BC. If these approaches demonstrate sufficiently concordant results to tissue-based testing, blood draws may quickly become a viable alternative to invasive biopsies.

In a cross-sectional study, 120 consecutive individuals from study centers in Ontario, who present with highly suspicious BC distant metastases who undergo biopsy to confirm BC recurrence will be enrolled (enrollment will be continued until 100 subjects with confirmed metastatic breast cancer have been enrolled). Blood samples for the circulating factors will be taken within 30 days prior to the tissue biopsy. Patient and tumor characteristics will be recorded. At the end of study, liquid biopsy (CTCs and ctDNA) analyses will be performed blinded to biopsy results. Investigators will continuously review the number of participants in each BC subtype. Cases with tissue biopsy results not classified as definite or highly suspicious for metastatic breast cancer by the treating physician will be re-assessed after six month of study entry in an attempt to classify them as having metastatic breast cancer or not. This aims to confirm/rule out breast cancer or other diagnosis.

The overall anticipated public and/or scientific benefit of the study is to demonstrate the concordance between liquid (blood) biopsy and tissue based tests in terms of the presence of cancer cells, hormone receptors, HER2 status etc. so these tests could be used in the future to confirm diagnosis using a non-invasive procedure. The results of this study will advance our understanding of liquid biomarkers and ideally improve the care journey for breast cancer patients by not subjecting them to invasive and potentially dangerous biopsy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years of age) diagnosed with primary breast cancer (BC) any subtype ER/PgR+ and HER2, triple negative or HER2+ at least 6 months before suspected metastases were identified
* Patients must have suspected recurrent metastatic BC that will be confirmed by tissue biopsy that is expected to yield tissue adequate for histologic examination (sampling expected to yield material for cytologic evaluation only does not satisfy this criterion)
* The suspected metastases must be outside the ipsilateral breast, axilla infra/supraclavicular areas. In those with suspected metastases in contralateral axilla, infra/supraclavicular areas only a new contralateral breast primary must be excluded by physical exam, mammogram and MRI

Exclusion Criteria:

* Only locoregional recurrence (ipsilateral breast, axilla, infra/supraclavicular) suspected (see above regarding potential contralateral axillary or infra/supraclavicular metastases as only site of metastasis)
* Tissue biopsy occurs prior to blood collection for CTCs and ctDNA
* New treatment for suspected metastases commences prior to blood collection for CTCs and ctDNA
* Patient has received previous lines of systemic treatment for metastatic BC
* Previous history of an invasive non-BC apart from cancers treated with curative intent at least 5 years previously with no recurrence since diagnosis, with the exception of a non-melanoma skin cancer
* Patients unable or unwilling to undergo a tissue biopsy
* Patients unable to provide informed consent
* Patients undergoing only cytologic evaluation of suspected metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study cohort will be selected from the Breast Cancer patients visiting London Regional Cancer Program for the treatment of their disease.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Concordance between liquid and tissue biopsy in terms of presence or absence of Cancer | Its a single visit study and the study investigators try to have a blood draw from patients within 30 days prior to tissue biopsy.
  To analyze concordance between liquid biopsy, CTCs (Epic Sciences) and ctDNA (academic assays based on mutations and/or epigenetic changes), with biopsy results (presence or absence of cancer), and with all blood assays being conducted blinded to tissue biopsy results

SECONDARY OUTCOMES:
Concordance between liquid and tissue biopsy in terms of hormone and HER2 status | Its a single visit study and study investigators try to have a blood draw from patients within 30 days prior to tissue biopsy.
  To conduct secondary analyses of the concordance between hormone receptor and HER2 status identified on tissue specimens with those identified on CTCs (Epic Sciences).
Classification of tissue biopsy results | Its a single visit study and study investigators try to have a blood draw from patients within 30 days prior to tissue biopsy.
  To classify tissue biopsy results according to the interpretation of the local pathologist, the treating physician (primary comparator) and the study investigators (interpretations to include clinical data such as physical exam, radiologic investigations, blood work as available).
Exploratory analysis | Its a single visit study and study investigators try to have a blood draw from patients within 30 days prior to tissue biopsy.
  To conduct exploratory analyses of the associations between tumor markers and CTCs or ctDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Lohmann, MD, PhD, Principal Investigator — London Regional Cancer Program
Locations (1):
- London Regional Cancer Program, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Simmons C, Miller N, Geddie W, Gianfelice D, Oldfield M, Dranitsaris G, Clemons MJ. Does confirmatory tumor biopsy alter the management of breast cancer patients with distant metastases? Ann Oncol. 2009 Sep;20(9):1499-1504. doi: 10.1093/annonc/mdp028. Epub 2009 Mar 18. PMID 19299408
- [Result] Macfarlane R, Seal M, Speers C, Woods R, Masoudi H, Aparicio S, Chia SK. Molecular alterations between the primary breast cancer and the subsequent locoregional/metastatic tumor. Oncologist. 2012;17(2):172-8. doi: 10.1634/theoncologist.2011-0127. Epub 2012 Jan 20. PMID 22267852
- [Result] Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med. 2004 Aug 19;351(8):781-91. doi: 10.1056/NEJMoa040766. PMID 15317891
- [Result] Paoletti C, Muniz MC, Thomas DG, Griffith KA, Kidwell KM, Tokudome N, Brown ME, Aung K, Miller MC, Blossom DL, Schott AF, Henry NL, Rae JM, Connelly MC, Chianese DA, Hayes DF. Development of circulating tumor cell-endocrine therapy index in patients with hormone receptor-positive breast cancer. Clin Cancer Res. 2015 Jun 1;21(11):2487-98. doi: 10.1158/1078-0432.CCR-14-1913. Epub 2014 Nov 7. PMID 25381338
- [Result] Fujii T, Reuben JM, Huo L, Espinosa Fernandez JR, Gong Y, Krupa R, Suraneni MV, Graf RP, Lee J, Greene S, Rodriguez A, Dugan L, Louw J, Lim B, Barcenas CH, Marx AN, Tripathy D, Wang Y, Landers M, Dittamore R, Ueno NT. Androgen receptor expression on circulating tumor cells in metastatic breast cancer. PLoS One. 2017 Sep 28;12(9):e0185231. doi: 10.1371/journal.pone.0185231. eCollection 2017. PMID 28957377
- [Result] Scher HI, Graf RP, Schreiber NA, McLaughlin B, Lu D, Louw J, Danila DC, Dugan L, Johnson A, Heller G, Fleisher M, Dittamore R. Nuclear-specific AR-V7 Protein Localization is Necessary to Guide Treatment Selection in Metastatic Castration-resistant Prostate Cancer. Eur Urol. 2017 Jun;71(6):874-882. doi: 10.1016/j.eururo.2016.11.024. Epub 2016 Dec 12. PMID 27979426
- [Result] Meng S, Tripathy D, Frenkel EP, Shete S, Naftalis EZ, Huth JF, Beitsch PD, Leitch M, Hoover S, Euhus D, Haley B, Morrison L, Fleming TP, Herlyn D, Terstappen LW, Fehm T, Tucker TF, Lane N, Wang J, Uhr JW. Circulating tumor cells in patients with breast cancer dormancy. Clin Cancer Res. 2004 Dec 15;10(24):8152-62. doi: 10.1158/1078-0432.CCR-04-1110. PMID 15623589
- [Result] Janni WJ, Rack B, Terstappen LW, Pierga JY, Taran FA, Fehm T, Hall C, de Groot MR, Bidard FC, Friedl TW, Fasching PA, Brucker SY, Pantel K, Lucci A. Pooled Analysis of the Prognostic Relevance of Circulating Tumor Cells in Primary Breast Cancer. Clin Cancer Res. 2016 May 15;22(10):2583-93. doi: 10.1158/1078-0432.CCR-15-1603. Epub 2016 Jan 5. PMID 26733614
- [Result] Coombes RC, Page K, Salari R, Hastings RK, Armstrong A, Ahmed S, Ali S, Cleator S, Kenny L, Stebbing J, Rutherford M, Sethi H, Boydell A, Swenerton R, Fernandez-Garcia D, Gleason KLT, Goddard K, Guttery DS, Assaf ZJ, Wu HT, Natarajan P, Moore DA, Primrose L, Dashner S, Tin AS, Balcioglu M, Srinivasan R, Shchegrova SV, Olson A, Hafez D, Billings P, Aleshin A, Rehman F, Toghill BJ, Hills A, Louie MC, Lin CJ, Zimmermann BG, Shaw JA. Personalized Detection of Circulating Tumor DNA Antedates Breast Cancer Metastatic Recurrence. Clin Cancer Res. 2019 Jul 15;25(14):4255-4263. doi: 10.1158/1078-0432.CCR-18-3663. Epub 2019 Apr 16. PMID 30992300
- [Result] Bratman SV, Newman AM, Alizadeh AA, Diehn M. Potential clinical utility of ultrasensitive circulating tumor DNA detection with CAPP-Seq. Expert Rev Mol Diagn. 2015 Jun;15(6):715-9. doi: 10.1586/14737159.2015.1019476. Epub 2015 Mar 16. PMID 25773944
- [Result] Newman AM, Lovejoy AF, Klass DM, Kurtz DM, Chabon JJ, Scherer F, Stehr H, Liu CL, Bratman SV, Say C, Zhou L, Carter JN, West RB, Sledge GW, Shrager JB, Loo BW Jr, Neal JW, Wakelee HA, Diehn M, Alizadeh AA. Integrated digital error suppression for improved detection of circulating tumor DNA. Nat Biotechnol. 2016 May;34(5):547-555. doi: 10.1038/nbt.3520. Epub 2016 Mar 28. PMID 27018799
- [Result] Visvanathan K, Fackler MS, Zhang Z, Lopez-Bujanda ZA, Jeter SC, Sokoll LJ, Garrett-Mayer E, Cope LM, Umbricht CB, Euhus DM, Forero A, Storniolo AM, Nanda R, Lin NU, Carey LA, Ingle JN, Sukumar S, Wolff AC. Monitoring of Serum DNA Methylation as an Early Independent Marker of Response and Survival in Metastatic Breast Cancer: TBCRC 005 Prospective Biomarker Study. J Clin Oncol. 2017 Mar;35(7):751-758. doi: 10.1200/JCO.2015.66.2080. Epub 2016 Nov 21. PMID 27870562
- [Result] Shen SY, Singhania R, Fehringer G, Chakravarthy A, Roehrl MHA, Chadwick D, Zuzarte PC, Borgida A, Wang TT, Li T, Kis O, Zhao Z, Spreafico A, Medina TDS, Wang Y, Roulois D, Ettayebi I, Chen Z, Chow S, Murphy T, Arruda A, O'Kane GM, Liu J, Mansour M, McPherson JD, O'Brien C, Leighl N, Bedard PL, Fleshner N, Liu G, Minden MD, Gallinger S, Goldenberg A, Pugh TJ, Hoffman MM, Bratman SV, Hung RJ, De Carvalho DD. Sensitive tumour detection and classification using plasma cell-free DNA methylomes. Nature. 2018 Nov;563(7732):579-583. doi: 10.1038/s41586-018-0703-0. Epub 2018 Nov 14. PMID 30429608
- [Result] Shen SY, Burgener JM, Bratman SV, De Carvalho DD. Preparation of cfMeDIP-seq libraries for methylome profiling of plasma cell-free DNA. Nat Protoc. 2019 Oct;14(10):2749-2780. doi: 10.1038/s41596-019-0202-2. Epub 2019 Aug 30. PMID 31471598
- [Result] Gion M, Peloso L, Mione R, Vignati G, Fortunato A, Saracchini S, Biasioli R, Gulisano M, Cappelli G. Tumor markers in breast cancer monitoring should be scheduled according to initial stage and follow-up time: a prospective study on 859 patients. Cancer J. 2001 May-Jun;7(3):181-90. PMID 11419026
- [Result] Mariani L, Miceli R, Michilin S, Gion M. Serial determination of CEA and CA 15.3 in breast cancer follow-up: an assessment of their diagnostic accuracy for the detection of tumour recurrences. Biomarkers. 2009 Mar;14(2):130-6. doi: 10.1080/13547500902770090. PMID 19330591